CLINICAL TRIAL: NCT03378141
Title: Evaluate a Feasibility Study of Integrating Maternal Nutrition Interventions in Existing Reproductive, Maternal, Newborn and Child Health Services in Uttar Pradesh, India
Brief Title: Maternal Nutrition Interventions in Uttar Pradesh, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-09-11
Record Dates: First submitted 2017-10-09; First posted 2017-12-19 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Anemia; Undernutrition; Underweight; Stunting; Maternal Malnutrition
MeSH Terms: conditions — Anemia; Malnutrition; Thinness; Growth Disorders

STUDY DESIGN:
Intervention Model Description: * The impact evaluation follows a cluster randomized controlled trial design with repeated cross-sectional surveys at baseline and endline
  * The nested cohort study follows a prospective randomized controlled design (embedded in overall impact evaluation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A&T- intensive (Experimental): A&T-intensive arm receive standard MNCH services and intensified maternal nutrition behavior change intervention. Intervention includes provision of IFA and calcium supplements, interpersonal counseling on diet during pregnancy and consumption of IFA and calcium, community mobilization, and adequate weight-gain monitoring during pregnancy
  Interventions: Behavioral: Maternal Nutrition Behavior change
- A&T-non intensive (No Intervention): A&T-non intensive arm only receives standard MNCH services

INTERVENTIONS:
Behavioral: Maternal Nutrition Behavior change — Counseling and community mobilization
  Arms: A&T- intensive

SUMMARY:
Maternal nutrition has been a long-standing concern of health authorities globally and in India. Despite the availability of proven, affordable interventions, and progressive policies and program platforms such as Maternal, Newborn and Child Health (MNCH) services, a streamlined package of proven maternal nutrition services is not reaching the majority of women during pregnancy.

Alive & Thrive India aims to test the feasibility of integrating a package of maternal nutrition interventions in routine Reproductive, Maternal, Newborn and Child Health (RMNCH) services.These include provision of IFA and calcium supplements, interpersonal counseling on diet during pregnancy and consumption of IFA and calcium, community mobilization, and adequate weight-gain monitoring during pregnancy.

This proposed evaluation aims to assess the feasibility of integrating maternal nutrition interventions into an existing RMNCH services in India, using a cluster-randomized evaluation design, complemented with a nested cohort study.

DETAILED DESCRIPTION:
Maternal nutrition has been a long-standing concern of health authorities globally and in India. Despite the availability of proven, affordable interventions, and progressive policies and program platforms such as Maternal, Newborn and Child Health (MNCH) services, a streamlined package of proven maternal nutrition services is not reaching the majority of women during pregnancy. This undermines national efforts to improve maternal and newborn survival; and reduce morbidity, malnutrition and disabilities in women and children.

Reducing maternal and child mortality are the most important goals of the National Health Mission with major strategic investments being made by Government of India to achieve these goals. The Maternal Mortality Ratio in India has shown a considerable decline from 424/100,000 live births in 1992-1993 to 167 in 2010-2013. These maternal deaths are exacerbated by the high burden of malnutrition and poor dietary intakes during and before pregnancy. The same nutritional deficits also contribute to low birth weight that in turn, is associated with higher infant mortality (which is at 37 per 1,000 live birth in 2015. Anemia remains a significant public health problem in India, affecting 53% women of reproductive age and 50% pregnant women, with a minimal decline during the last decade. Further more, nearly a third of women and 44.7% of girls aged 15 to 18 years have a low body mass index (BMI less than 18.5), thus entering pregnancy in a vulnerable state. During pregnancy, on average, women gained only 7 kg, much lower than the recommended weight gain of 10-12 kg.

In 2016, the World Health Organization (WHO) issued new guidelines on antenatal care (ANC) for a positive pregnancy experience to improve nutrition through dietary interventions and micronutrient supplements, along with health system interventions to improve the utilization and quality of ANC. Indian policy framework includes food supplementation, iron and folic acid (IFA) and calcium supplementation to improve maternal nutrition. In addition, with the advent of the National Health Mission in 2006, the Reproductive, Maternal, Newborn and Child Health (RMNCH) gained priority and investments were made to expand the quality and coverage of maternal health services, including ANC contacts.

Despite policy guidance, the nutrition content of ANC (e.g. IFA and calcium supplementation, monitoring and counseling on weight gain) remains to be prioritized. According to the National Family and Health Survey 2015-2016 (NFHS-4), nearly 90% of pregnancies in India were registered for health services, 51% received at least 4 ANC visits, but only 30% reported consuming 100 or more IFA tablets during their last pregnancy. In Uttar Pradesh, the proportion of women who received at least 4 ANC visits increased from 11% to 26% during the last decade. However, the proportion of women consuming IFA supplements more than doubled (6% to 13%) but is still very low. This suggests that there is a need to fully utilize the existing contacts to deliver maternal nutrition interventions within MNCH services.

Alive & Thrive (A&T) supports scaling up of nutrition interventions to save lives, prevent illnesses, and contributes to healthy growth and development through improved maternal nutrition, breastfeeding and complementary feeding in several countries. In India, A&T aims to test the feasibility of integrating a package of maternal nutrition interventions that align with the latest global evidence and the national policies and guidelines of Government of India within routine RMNCH services. These include provision of IFA and calcium supplements, interpersonal counseling on diet during pregnancy and consumption of IFA and calcium, community mobilization, and adequate weight-gain monitoring during pregnancy.

The primary objectives of the proposed evaluation are to answer the following questions using a cluster-randomized evaluation design:

* Can the coverage and utilization of key maternal nutrition interventions be improved by integrating nutrition-focused social behavior change communication (SBC) and systems strengthening approaches into ANC services under RMNCH program?
* What factors affect effective integration of maternal nutrition interventions into a well-established government ANC service delivery platform under RMNCH program?
* What are the impacts of program on: 1) consumption of diversified foods and adequate intake of micronutrient, protein and energy compared to recommended intake; 2) intake of IFA and calcium supplements during pregnancy; 3) weight gain monitoring; and 4) early initiation of breastfeeding.

In addition, a nested cohort will be conducted to complement the overall impact evaluation with the following primary objectives:

* To collect objective measures of maternal nutrition outcomes such as weight gain during pregnancy, anemia, IFA and calcium consumption, and diet diversity and adequate intake (including macro- and micro-nutrient intakes).
* To understand the key barriers/facilitators which influence intentions and practices related to maternal nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Recently delivered women with children <6 months of age
* Pregnant women in first, second and third trimester
* Husbands of these women
* Mothers or mother-in-law of these women
* Frontline health workers in the areas

Exclusion Criteria:

* Age <18
* Mental health problems that make it difficult for the respondent to answer the questions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Use of iron-folic acid and calcium supplements | During pregnancy (about 9 months) and up to 24 weeks postpartum
  Recall the total number of IFA and calcium tablets consumed throughout the last pregnancy
Dietary diversity during pregnancy | During pregnancy (about 9 months)
  Number of food groups women consumed and proportion of women consumed at least 5 food groups

SECONDARY OUTCOMES:
Coverage of maternal nutrition intervention | During pregnancy (about 9 months) and up to 24 weeks postpartum
  The proportion of pregnant and recently delivery women expose to and use of maternal nutrition intervention during the last 2 year
Micronutrient adequacy of the diet | During pregnancy (about 9 months)
  Dietary intakes of 11 vitamins and micronutrients
Weight gain monitoring during pregnancy | During pregnancy (about 9 months)
  proportion of women who are weighed and counselled about adequate weight gain and the numbers time women are weighed
Early initiation of breastfeeding | Infants up to 6 months
  The proportion of newborns aged less than 6 months who were breastfed within 1 hour of birth
Exclusive breastfeeding | Infants up to 6 months
  The proportion of infants aged less than 6 months who were exclusively breastfed on the day preceding the interview
Anemia (Hb levels) | During pregnancy (about 9 months) and up to 24 weeks postpartum
  The proportion of pregnant and recently delivered women diagnosed with moderate or severe anemia

CONTACTS AND LOCATIONS:
Overall Officials: Phuong H Nguyen, Principal Investigator — International Food Policy Research Institute
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Young MF, Bootwala A, Kachwaha S, Avula R, Ghosh S, Sharma PK, Shastri VD, Forissier T, Menon P, Nguyen PH. Understanding Implementation and Improving Nutrition Interventions: Barriers and Facilitators of Using Data Strategically to Inform the Implementation of Maternal Nutrition in Uttar Pradesh, India. Curr Dev Nutr. 2021 Jun 2;5(6):nzab081. doi: 10.1093/cdn/nzab081. eCollection 2021 Jun. PMID 34222761
- [Derived] Nguyen PH, Kachwaha S, Tran LM, Avula R, Young MF, Ghosh S, Sharma PK, Escobar-Alegria J, Forissier T, Patil S, Frongillo EA, Menon P. Strengthening Nutrition Interventions in Antenatal Care Services Affects Dietary Intake, Micronutrient Intake, Gestational Weight Gain, and Breastfeeding in Uttar Pradesh, India: Results of a Cluster-Randomized Program Evaluation. J Nutr. 2021 Aug 7;151(8):2282-2295. doi: 10.1093/jn/nxab131. PMID 34038529
- [Derived] Nguyen PH, Martin-Prevel Y, Moursi M, Tran LM, Menon P, Ruel MT, Arimond M. Assessing Dietary Diversity in Pregnant Women: Relative Validity of the List-Based and Open Recall Methods. Curr Dev Nutr. 2019 Nov 18;4(1):nzz134. doi: 10.1093/cdn/nzz134. eCollection 2020 Jan. PMID 32258987